CLINICAL TRIAL: NCT05823714
Title: Venetoclax + Azacytidine Followed by Modified BUCY Conditioning Regimen for High-risk Myelodysplastic Syndromes (MDS) and High-risk or Relapsed/Refractory Acute Myeloid Leukemia (AML) Undergoing Allogeneic Hematopoietic Stem Cell Transplantation (Allo-HSCT)
Brief Title: Venetoclax+Azacytidine+Modified BUCY Conditioning Regimen for Acute Myeloid Leukemia and Myelodysplastic Syndromes Undergoing Allo-HSCT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VA+mBUCY-01
Record Dates: First submitted 2023-02-27; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-02

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplantation; Acute Myeloid Leukemia; Myelodysplastic Syndrome
Keywords: venetoclax; azacytidine; hematopoietic stem cell transplantation; acute myeloid leukemia; myelodysplastic syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VEN+AZA+Modified BUCY (Experimental)
  Interventions: Drug: VEN+AZA+Modified BUCY

INTERVENTIONS:
Drug: VEN+AZA+Modified BUCY — Venetoclax: 200mg/day*7days（It should be combined with triazole antifungal drugs).
  Azacytidine: 75mg/ m²/day*7days.

SUMMARY:
The purpose of this prospective, open-label, single-center study is to evaluate the efficacy and safety of VEN-AZA (venetoclax and azacytidine) followed by modified BUCY (busulfan and cyclophosphamide) as conditioning regimen for high-risk myelodysplastic syndrome (MDS) and high-risk or relapsed/refractory acute myeloid leukemia (AML) undergoing allogeneic hematopoietic stem cell transplantation (allo-HSCT).

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (Allo-HSCT) is the only potentially curative therapy for patients with myelodysplastic syndrome (MDS) and acute myeloid leukemia (AML). However, relapse remains a leading cause for treatment failure after hematopoietic cell transplantation (HCT) in patients, optimization of conditioning regimen can improve prognosis and decrease relapse. Abnormal gene methylation is common in AML and MDS patients. Azacytidine is a DNA methylation transferase inhibitor that can re-express tumor suppressor genes in leukemia cells. Venetoclax is a selective BCL-2 inhibitor, which has antitumor activity against a variety of hematological malignancies. The combination of the two drugs show a synergistic anti-tumor effect. The objective of this study is to evaluate the safety and efficacy of VEN-AZA regimen followed by Allo-HSCT in the treatment of high-risk MDS and high-risk or relapsed/refractory AML.

ELIGIBILITY:
Inclusion Criteria:

1. Age 8 to 65 years;
2. Diseases must be MDS and AML; high-risk MDS: int-2 risk, high risk by the IPSS; IPSS-R int-risk (> 3.5 points), high risk, very high risk; high risk,very high risk by the WPSS; high-risk or relapsed/refractory AML: (1) age≥60 years; (2) High white blood cell count at first diagnosis (WBC≥100*10^9/L); (3) secondary AML (previous history of MDS, myeloproliferative disease, or treatment-related AML, etc.); (4) Complicated with extramedullary leukemia, such as central nervous system leukemia, granulocytic sarcoma, hepatosenomegaly; （5）high risk factors and relapsed/refractory AML（reference 2022-AML-ELN guideline）（6）not in remission or ≥CR2 before transplantation;
3. Must need a bone marrow transplant;
4. Must have the ability to observe the efficacy and events;
5. Patient must have ability to understand and willingness to provide written informed consent prior to participation in the study and any related procedures being performed.

Exclusion Criteria:

1. Age <8 or >65 years;
2. Uncontrolled bacterial, viral, fungal, or other infection before conditioning regimen;
3. Pregnant or lactating females;
4. Current participation in another clinical trial;
5. Contra-indication to one of the drug of the regimen;
6. Any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver or other organ system that may place the patient at undue risk to undergo the agents included in the conditioning regimen.

Ages: 8 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2025-01-20 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
disease-free survival (DFS) | 3 years after transplantation
  It is measured from the time from randomization to the first of relapse or death.
overall survival (OS) | 3 years after transplantation
  It is measured from the time of entry into this trial to the date of death from any cause; patients not known to have died at last follow-up are censored on the date they were last known to be alive.

SECONDARY OUTCOMES:
veno-occlusive disease (VOD) | 3 years after transplantation
  incidence of veno-occlusive disease (VOD) events (refer to modified Seattle Criteria of VOD)
graft-versus-host disease (GvHD) | 3 years after transplantation
  incidence and severity of acute (aGvHD) and chronic graft-versus-host disease (cGvHD) (aGvHD refer to Glucksberg Criteria and cGvHD refer to the National Institutes of Health Consensus)
transplant related mortality (TRM) | 3 years after transplantation
  cumulative incidence of transplant related mortality
Regimen related toxicity | 3 years after transplantation
  Number of participants with conditioning regimen related toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Depei Wu Wu, MD, Study Chair — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China